CLINICAL TRIAL: NCT04539821
Title: Virtual Pain Care for High Risk Veterans on Opioids During COVID19 (and Beyond)
Brief Title: Virtual Pain Care Management (COVID-19)
Acronym: VCPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: C19 20-397; NCT04228250 (obsolete NCT alias)
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain
Keywords: buprenorphine
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This single-arm feasibility study will be conducted in two VA sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VCPM (Other): VCPM is a multi-component intervention consisting of already-established care processes and materials. First, the patient is mailed or emailed (based on their preference) an informational packet prior to intake appointment. Second, using the collaborative medication management model established in VHA,3 the intake appointment is led by the CPS using a standardized intake evaluation. The CPS and physician design a plan presented to the patient. If BUP switch is offered and accepted, the physician completes additional brief evaluations, including a history, medication review, treatment planning, and discussion of other VCPM components, using two-way audio-video visits (with telephone as a back-up).
  Interventions: Other: VCPM

INTERVENTIONS:
Other: VCPM — VCPM is a multi-component intervention consisting of already-established care processes and materials.
  Other Names: Virtual Chronic Pain Management

SUMMARY:
The COVID-19 pandemic is exacerbating the challenges faced by Veterans at risk of opioid overdose including Veterans prescribed moderate-to-high dose long-term opioid therapy (LTOT) whose usual treatment resources and coping strategies may be inaccessible. This project combines established VA care components to deploy and evaluate virtual models of care for Veterans on high-risk LTOT to meet the dual challenges of maintaining social distancing and delivery high quality care.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must currently receive LTOT for chronic pain at 50 mg morphine equivalent daily dose

Exclusion Criteria:

Exclusion criteria at baseline are:

* dementia diagnosis or moderate-severe cognitive impairment
* unstable or severe untreated psychiatric disorder or medical disease that requires hospitalization
* documentation of suspected controlled substance diversion
* inability to communicate by phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Adams Moore, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: for this single arm all participants receive VCPM
Period: Overall Study
Arm/Group | Single Arm
Started | 44
Engaged in CPS Care (these individuals engaged in care with the clinical pharmacists and made changes to their opioid regimen) | 21
Completed | 19
Not Completed | 25
Not completed — Withdrawal by Subject | 2
Not completed — continued care with their physician | 20
Not completed — treatment needs outside scope of VCPM | 3

BASELINE CHARACTERISTICS:
Groups:
- VCPN Single Arm: for this single arm all participants receive VCPM
Arm/Group | VCPN Single Arm
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 38
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Agree to Change in Their Opioid Regimen, Including Buprenorphine Transfer
Description: Using shared decision-making with Veterans, we will based the measure on clinical reports of patient change in opioid regimen. This would be tapering (reducing opioid dose), discontinuation, or transfer to buprenorphine. Any reduction or change was considered positive for change, even if the patients returned to their initial dose. The number of patients who agree to change their opioid regimen provides a realistic indicator of overall feasibility/acceptability.
Time Frame: 30 days
Population: All participants who completed the initial CPS visit
Measure: Count of Participants; unit: Participants
Arm/Group | VCPM
Number analyzed (Participants) | 44
Participants | 19

2. Secondary Outcome: Number of Participants Retained in Care at End of Study
Description: Of participants who engaged in initial treatment the number who completed or were retained in care at the end of the study provides a outcome measure of engagement
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | VCPM
Number analyzed (Participants) | 19
participants | 17

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | VCPM
All-Cause Mortality (participants affected / at risk) | 1/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 2/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VCPM (N=44)
Discontinuation of Buprenorphine (Gastrointestinal disorders) | 2 (2) — expected side effects of Buprenorphine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT04539821/Prot_SAP_000.pdf